CLINICAL TRIAL: NCT02921711
Title: TRAIL: Treatment of Intracranial Aneurysms With LVIS® System
Acronym: TRAIL
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRAIL
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LVIS®
  Interventions: Device: LVIS®

INTERVENTIONS:
Device: LVIS® — Low-profile Visualized Intraluminal Support device

SUMMARY:
A prospective, multicenter, observational assessment of the safety and effectiveness of the LVIS® device in the treatment of wide necked intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or patient's legally authorized representative has been informed about the confidentiality of the study and has agreed to the collection of his/her personal data
2. Patient has a ruptured or unruptured intracranial aneurysm for which:

   * The parent artery has a diameter ≥ 2.0mm and ≤ 4.5 mm;
   * The aneurysm neck size is ≥ 4mm or its dome-to-neck ratio is < 2 (wide neck)
   * Endovascular treatment with coils and one or more LVIS® devices has been determined necessary for the patient by the multidisciplinary team
3. Patient is aged ≥ 18 years
4. Patient presents with a WFNS score between 0 and 3
5. Patient has agreed to attend follow-up appointments

Exclusion Criteria:

1. The use of an endovascular stent other than LVIS® has been determined necessary
2. Patient presents with medical or surgical co-morbidities limiting his/her life expectancy to less than one year
3. Patient has a contraindication to platelet inhibition treatment
4. Patient requires retreatment of an aneurysm previously treated with a stent
5. Patient is pregnant
6. Patient has multiple aneurysms to be treated in one procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged minimum of 18 years with an intracranial aneurysm in whom stent-assisted coiling has been determined to be the appropriate treatment strategy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Anatomical stability of aneurysm treatment compared to the initial occlusion rate of the aneurysm | 6 months
Anatomical stability of aneurysm treatment compared to the initial occlusion rate of the aneurysm | 18 months
Retreatment rate | 6 months
Retreatment rate | 18 months
Morbidity rate | 6 months
Morbidity rate | 18 months
Mortality rate | 6 months
Mortality rate | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Mounayer, Prof., Principal Investigator — CHU Limoges; Limoges, France; Michel Piotin, M.D., Principal Investigator — Fondation Rothschild; Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Safety and effectiveness of the Low Profile Visualized Intraluminal Support (LVIS and LVIS Jr) devices in the endovascular treatment of intracranial aneurysms: results of the TRAIL multicenter observational study — https://pubmed.ncbi.nlm.nih.gov/29175829/